CLINICAL TRIAL: NCT04352192
Title: The Effect of Kinesiotaping on Bioelectrical Muscle Activity
Brief Title: Effect of Kinesiotaping on Muscle Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assistant professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: hdenizkulli4
Record Dates: First submitted 2020-04-08; First posted 2020-04-20 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: kinesiotaping; EMG

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping Group (Experimental): The group in which kinesiotaping is going to be applied to biceps brachii muscle of participants and will assess EMG activities before KT, immediately after KT, after 30 minutes and 24 hours of KT. The EMG analysis will be performed during maximum isometric voluntary contraction of biceps brachii muscle.
  Interventions: Other: Kinesiotaping
- Control Group (No Intervention): The group in which kinesiotaping is not going to be applied. EMG activities will be assessed first assessment and after 10th minutes, 30th minutes and 24th hours of the first assessment. The EMG analysis will be performed during maximum isometric voluntary contraction of biceps brachii muscle.

INTERVENTIONS:
Other: Kinesiotaping — For kinesiotaping, the elbow positioned in 30°-45° flexion and kinesiotaping facilitation technique is applied origin to insertion of biceps brachii muscle.
  Arms: Kinesiotaping Group

SUMMARY:
The aim of the investigator's study is to analyze the effect of kinesiotaping (KT) on the electrical activity of the muscle by using time and frequency domain analysis of the electromyography (EMG) signals.

DETAILED DESCRIPTION:
The kinesiotaping (KT) is a taping technique that is commonly used to improve muscle performance and facilitate or inhibit muscle activity in rehabilitation. A study reported that KT application did not change electrical activity in the early period (immediately after KT, 5th and 10 minutes after KT). However, another study showed that EMG activity increased 24 hours after KT application. A study revealed that the KT produced more EMG activity compare to placebo taping. In conclusion, the effect of KT on electrical muscular activity was arguable in the literature.

ELIGIBILITY:
Inclusion Criteria:

* To be right-handed-dominant
* To have normal or corrected vision
* To have no formal history of any resistance training.

Exclusion Criteria:

* To have history of neurological or recent musculoskeletal injury

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
The first assessment of electromyographic activity | at inclusion
  The electromyographic activity of biceps brachii muscle will be measured during elbow maximum isometric flexion by using electromyography device before KT for KT group or as a first assessment of the control group. The test will be repeated three times.
The second assessment of electromyographic activity | after KT application for KT group or at 10th minutes after the first assessment
  The electromyographic activity of biceps brachii muscle will be measured during elbow maximum isometric flexion by using electromyography device immediately after KT application for KT group or at 10th minutes after the first assessment as a second assessment of the control group. The test will be repeated three times.
The third assessment of electromyographic activity | 30 minutes after the second assessment
  The electromyographic activity of biceps brachii muscle will be measured during elbow maximum isometric flexion by using electromyography device at 30 minutes after the second assessment. The test will be repeated three times.
The last assessment of electromyographic activity | at 24 hours after KT application or the second assessment
  The electromyographic activity of biceps brachii muscle will be measured during elbow maximum isometric flexion by using electromyography device at 24 hours after KT application or the second assessment. The test will be repeated three times.

SECONDARY OUTCOMES:
The first assessment of maximum isometric voluntary contraction torque | at inclusion
  The produced elbow flexion torque during first EMG assessment will be recorded at 90° elbow flexion using isokinetic dynamometer.
The second assessment of maximum isometric voluntary contraction torque | after KT application for KT group or at 10th minutes after the first assessment
  The produced elbow flexion torque during second EMG assessment will be recorded at 90° elbow flexion using isokinetic dynamometer.
The third assessment of maximum isometric voluntary contraction torque | 30 minutes after the second assessment
  The produced elbow flexion torque during third EMG assessment will be recorded at 90° elbow flexion using isokinetic dynamometer.
The last assessment of maximum isometric voluntary contraction torque | at 24 hours after KT application or the second assessment
  The produced elbow flexion torque during the last EMG assessment will be recorded at 90° elbow flexion using isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal DENIZOGLU KULLI, PhD, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denizoglu Kulli H, Karabulut D, Arslan YZ. The prolonged effect of Kinesio Taping on joint torque and muscle activity. Somatosens Mot Res. 2023 Mar;40(1):39-45. doi: 10.1080/08990220.2022.2157394. Epub 2022 Dec 20. PMID 36538392